CLINICAL TRIAL: NCT06930235
Title: Effectiveness of Midodrine as an Adjuvant to Norepinephrine in Weaning Critically Ill Patients From Vasopressors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Khalaf Elsayed, Resident, Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-3-06MS
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Weaning critically ill patients from norepinephrine using midodrine as an adjuvant to norepinephrine (Active Comparator): Patients in group I will receive midodrine (10 mg orally every 8 hours) in addition to administered concurrently with ongoing intravenous norepinephrine after being on norepinephrine for more than 24 h.
  Interventions: Drug: Weaning critically ill patients from norepinephrine using midodrine as an adjuvant to norepinephrine
- Weaning critically ill patients from norepinephrine without use of midodrine as an adjuvant (Active Comparator): Patients in group II with ongoing intravenous norepinephrine only
  Interventions: Drug: Weaning critically ill patients from norepinephrine without use of midodrine as an adjuvant

INTERVENTIONS:
Drug: Weaning critically ill patients from norepinephrine using midodrine as an adjuvant to norepinephrine — • Patients in group I will receive midodrine (10 mg orally every 8 hours) in addition to administered concurrently with ongoing intravenous norepinephrine after being on norepinephrine for more than 24 hrs.
  Arms: Weaning critically ill patients from norepinephrine using midodrine as an adjuvant to norepinephrine
Drug: Weaning critically ill patients from norepinephrine without use of midodrine as an adjuvant — Patients in group II with ongoing intravenous norepinephrine only
  Arms: Weaning critically ill patients from norepinephrine without use of midodrine as an adjuvant

SUMMARY:
This study aims to evaluate the effectiveness of midodrine as an adjuvant to norepinephrine in weaning critically ill patients from vasopressors

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory hypotension on an intravenous vasopressor for more than 24 h but deemed clinically stable.
* Patients on noradrenaline support <10 μg/min

Exclusion Criteria:

* Known allergy to midodrine.
* Severe shock state, as evidenced by multiple vasopressor infusions or high vasopressor requirement (i.e. noradrenaline >10 μg/min)
* Patients with severe organic heart disease (e.g., heart failure, sever aortic stenosis), pregnancy, thyrotoxicosis or pheochromocytoma.
* Those with no enteral route available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2025-10-13 (Estimated)

PRIMARY OUTCOMES:
follow up of critically ill patients on vasopressors | 48 hours
  time of weaning from intravenous vasopressor (norepinephrine)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Costa-Pinto R, Yong ZT, Yanase F, Young C, Brown A, Udy A, Young PJ, Eastwood G, Bellomo R. A pilot, feasibility, randomised controlled trial of midodrine as adjunctive vasopressor for low-dose vasopressor-dependent hypotension in intensive care patients: The MAVERIC study. J Crit Care. 2022 Feb;67:166-171. doi: 10.1016/j.jcrc.2021.11.004. Epub 2021 Nov 18. PMID 34801917
- [Background] Hammond DA, Smith MN, Peksa GD, Trivedi AP, Balk RA, Menich BE. Midodrine as an Adjuvant to Intravenous Vasopressor Agents in Adults With Resolving Shock: Systematic Review and Meta-Analysis. J Intensive Care Med. 2020 Nov;35(11):1209-1215. doi: 10.1177/0885066619843279. Epub 2019 Apr 28. PMID 31030630
- [Background] Hamed M, Elseidy SA, Elkheshen A, Maher J, Elmoghrabi A, Zaghloul A, Panakos A, Panaich S, Saad M, Elbadawi A. The Use of Midodrine as an Adjunctive Therapy to Liberate Patients from Intravenous Vasopressors: A Systematic Review and Meta-analysis of Randomized Controlled Studies. Cardiol Ther. 2023 Mar;12(1):185-195. doi: 10.1007/s40119-023-00301-0. Epub 2023 Jan 21. PMID 36670331